CLINICAL TRIAL: NCT06793735
Title: Effectiveness of Telerehabilitation Plus Virtual Reality App in Patients With Subjective Cognitive Decline, and Mild Cognitive Impairment
Brief Title: Effectiveness of TeleVR App in Cognitive Decline and MCI Patients
Acronym: TeleVR24
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Maria Grazia Maggio, Health Researcher, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TeleVR App_24; Current Research Funds 2024 (Other Grant/Funding Number: Ministry of Health, Italy)
Record Dates: First submitted 2025-01-17; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Dysfunction; Subjective Health; Mild Cognitive Impairment; Alzheimer Disease; Parkinson Disease
Keywords: Telerehabilitation; Virtual Reality (VR); Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD); Cognitive Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Parkinson Disease | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial (RCT), participants are assigned to one of two intervention groups:
  Experimental Group (EG): Participants will undergo a telerehabilitation program using two non-immersive Virtual Reality (VR) apps (NeuroNation and The Sims Mobile) on smartphones or tablets. The intervention aims to enhance cognitive and social cognition skills through interactive exercises conducted remotely.
  Active Control Group (aCG): Participants will follow a traditional cognitive rehabilitation program using paper-based exercises targeting similar cognitive and social domains.
  Key Model Details:
  Randomization: Participants are randomly assigned to either the experimental or control group using a block randomization method to ensure balance between groups.
  Blinding: Outcome assessors will be blinded to group assignments to reduce bias.
  Duration: Both groups will follow a 6-week intervention program, with assessments at baseline (T0), post-intervention (T1), and at a 3-month f
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will use a single-blind design, where outcome assessors will be blinded to group assignments to minimize bias during the evaluation of results.
  Participants: Not masked. Participants will be aware of their assigned intervention (Telerehabilitation with Virtual Reality or traditional paper-based rehabilitation).
  Healthcare Providers/Therapists: Not masked. Therapists guiding the telerehabilitation sessions or traditional rehabilitation tasks will be aware of the group assignments.
  Outcome Assessors: Masked. Neuropsychological assessments, EEG analysis, gait analysis, eye movement evaluations, and MRI data interpretation will be performed by independent assessors who will not have information about group allocation.
  This masking strategy ensures an objective and unbiased assessment of the study's primary and secondary outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-VR Group (Experimental): Participants in this arm will undergo a Telerehabilitation program using Virtual Reality (VR) apps. This intervention is designed to improve cognitive and social cognition skills through interactive, engaging exercises conducted remotely.
  Interventions: Device: Telerehabilitation with Virtual Reality
- Active Control Group (aCG) (Active Comparator): Participants in this arm will receive a traditional cognitive rehabilitation program using paper-based exercises. The intervention targets the same cognitive and social domains as the experimental group but uses conventional rehabilitation methods.
  Interventions: Other: Traditional Cognitive Rehabilitation

INTERVENTIONS:
Device: Telerehabilitation with Virtual Reality — Participants assigned to the experimental group will engage in a six-week telerehabilitation program utilizing two non-immersive Virtual Reality (VR) applications, NeuroNation and The Sims Mobile. These apps are designed to enhance cognitive performance and social cognition skills through interactive and scientifically validated exercises. NeuroNation focuses on improving memory, attention, reasoning speed, and mental flexibility, while The Sims Mobile engages participants in realistic social scenarios that challenge their empathy, communication, and problem-solving abilities. The intervention involves three 30-minute sessions per week, which participants will complete remotely using smartphones or tablets. Therapists will provide weekly virtual check-ins to monitor progress, address questions, and ensure adherence to the protocol. This program aims to create an engaging and accessible rehabilitation experience while promoting real-life application of cognitive and social skills improv
  Arms: Tele-VR Group
Other: Traditional Cognitive Rehabilitation — Participants in the control group will follow a traditional rehabilitation protocol that relies on paper-based cognitive exercises. This program targets cognitive domains such as attention, memory, and executive functions through tasks like puzzles, memory challenges, and problem-solving activities. The intervention also spans six weeks, with participants completing three 30-minute sessions per week. During an initial session, participants will receive all necessary materials and instructions for completing the exercises independently at home. Therapists will provide weekly remote support via phone or video to track progress and address any concerns. This conventional approach serves as a baseline for comparison with the innovative telerehabilitation method in the experimental group.
  Arms: Active Control Group (aCG)

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a telerehabilitation program combined with a virtual reality (VR) app in improving cognitive performance and social skills in patients with Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI).

The main questions it aims to answer are:

Can a VR telerehabilitation program improve cognitive functions and social skills in patients with SCD and MCI? Are there measurable changes in brain activity, eye movements, and gait patterns after the intervention? Researchers will compare telerehabilitation with a VR group (Experimental Group - EG) to a traditional paper-based cognitive rehabilitation group (Active Control Group - aCG) to determine which approach is more effective.

Participants will:

Undergo an initial assessment, including neurological exams, neuropsychological tests, brain MRI, EEG, eye movement analysis, and gait evaluation.

Participate in a 6-week intervention program:

EG: Use VR apps on smartphones/tablets at home, guided remotely by a therapist. aCG: Perform traditional cognitive exercises using paper-based tasks. Complete follow-up assessments immediately after the intervention and again after three months.

This study will help determine whether telerehabilitation with VR can provide measurable cognitive and social benefits, contributing to improved care strategies for individuals at risk of dementia.

DETAILED DESCRIPTION:
This clinical trial aims to assess the effectiveness of a telerehabilitation program combined with a virtual reality (VR) app in enhancing cognitive performance and social skills in individuals with Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI).

Study Rationale SCD and MCI are considered critical stages in identifying individuals at risk for dementia. Both conditions are associated with cognitive and social impairments, as well as neurophysiological changes observable through advanced neuroimaging and EEG markers. While traditional cognitive rehabilitation has shown benefits, emerging evidence suggests that telerehabilitation combined with VR may offer enhanced outcomes through its interactive, engaging, and scalable nature.

Primary Objective Evaluate the potential efficacy of a telerehabilitation plus VR intervention in improving cognitive performance and social cognition skills in patients with SCD and MCI.

Secondary Objectives Assess neurophysiological changes (EEG and MRI biomarkers) following the intervention.

Evaluate gait patterns and eye movement parameters. Investigate the usability and patient compliance of the VR app-based intervention.

Study Design Type: Randomized Clinical Trial (RCT) Duration: 6 weeks intervention, with follow-up assessments at baseline (T0), post-intervention (T1), and 3 months after intervention (T2).

Population: Individuals aged 40-80 with SCD or MCI (AD and PD subtypes).

Intervention Groups:

Experimental Group (EG): Participants will use two non-immersive VR apps ("NeuroNation" and "The Sims Mobile") on smartphones/tablets for cognitive and socio-emotional skill training. Training will occur 3 times per week, 30 minutes per session, guided remotely by therapists.

Active Control Group (aCG): Participants will follow a traditional cognitive rehabilitation program using paper-based exercises targeting cognitive domains.

Assessment Tools:

Neuropsychological Assessment: MMSE, MoCA, FAB, Stroop Test, RAVLT, Trail Making Test (TMT-A/B), and more.

Neurophysiological Assessment: EEG and MRI scans for brain activity and structural analysis.

Gait Analysis: Timed Up and Go (TUG) Test with BTS G-WALK®. Eye Movement Analysis: Using an eye-tracking system for fixation, saccades, antisaccades, and smooth pursuit eye movements.

Usability Assessment: System Usability Scale (SUS).

Expected Outcomes:

Improved cognitive and social cognition performance in the experimental group compared to the control group.

Observable changes in EEG and MRI biomarkers correlating with cognitive improvements.

Enhanced usability and acceptance of VR-based telerehabilitation tools among participants.

Significance of the Study:

This trial seeks to bridge the gap between traditional cognitive rehabilitation and innovative, scalable, and cost-effective digital health interventions. Positive outcomes could establish telerehabilitation with VR as a standard intervention for cognitive and social rehabilitation in at-risk populations.

The study adheres to ethical principles outlined in the Declaration of Helsinki, and informed consent will be obtained from all participants before enrollment

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with MCI (AD and PD) according to the criteria of the National Institute on Aging-Alzheimer's Association (NIA-AA, Albert et al., 2011)
* Subjects diagnosed with SCD according to diagnostic criteria proposed in research settings (Molinuevo et al., 2017)
* All enrolled subjects must be aged between 40 and 80 years and have at least 5 years of education

Exclusion Criteria:

* Presence of psychiatric disorders (major depression, psychosis, anxiety disorders)
* Presence of severe dementia
* History of cerebral ischemia
* Contraindications to brain MRI: pregnant women, pacemakers, non-latest-generation metal joint prostheses, electrodes, neurostimulators, or prostheses that may interfere with magnetic fields, unless there is a written statement of suitability from the specialist who performed the intervention

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance Improvement | The time frame for assessing cognitive performance improvement is at baseline (T0), immediately post-intervention (T1, after 6 weeks), and at follow-up (T2, 3 months after the intervention).
  The primary objective is to evaluate the effectiveness of the telerehabilitation program combined with Virtual Reality (VR) in improving global cognitive performance. This includes assessing domains such as memory, attention, and executive functioning in patients with Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI).
Social Cognition Enhancement | Social cognition improvements will be evaluated over the same time frame as cognitive performance: baseline (T0), post-intervention (T1, after 6 weeks), and follow-up (T2, 3 months after the intervention).
  Another key objective is to examine the impact of the telerehabilitation program on social cognition skills. This involves measuring improvements in empathy, Theory of Mind, and overall social interaction abilities, which are critical for maintaining functional independence and quality of life.

SECONDARY OUTCOMES:
Neurophysiological Changes | Neurophysiological changes will be assessed at baseline (T0) and immediately post-intervention (T1, after 6 weeks).
  A secondary objective is to investigate the neurophysiological changes associated with the intervention. This includes analyzing EEG parameters (such as changes in alpha, theta, and beta rhythms) and MRI biomarkers (like hippocampal connectivity) to understand the underlying mechanisms driving cognitive and social improvements.
Gait and Motor Function Improvement | Gait and motor function assessments will occur at baseline (T0) and post-intervention (T1, after 6 weeks).
  This objective focuses on evaluating changes in motor function and gait performance, assessed through the Timed Up and Go (TUG) test. The aim is to explore potential links between cognitive rehabilitation and cognitive-motor integration.

CONTACTS AND LOCATIONS:
Overall Officials: Rosso Salvatore Calabrò, MD,PhD, Study Director — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD related to primary and secondary outcome measures will be shared. This includes data on cognitive performance, social cognition, neurophysiological parameters (EEG and MRI biomarkers), gait analysis, and eye movement metrics. Data will be made available to qualified researchers upon reasonable request, following ethical and legal guidelines to ensure participant confidentiality. Access will be provided through a secure platform for a limited period after the study's completion. Specific requests will be evaluated on a case-by-case basis, and approved researchers must agree to terms of use.
Supporting Information: SAP
Time Frame: IPD and supporting documentation, including the Statistical Analysis Plan (SAP), will be available starting 6 months after the study's primary completion date. Access will be provided for 5 years from the initial availability date, ensuring adequate time for secondary analyses while maintaining relevance to ongoing research efforts.
Access Criteria: Requests for access to Individual Participant Data (IPD) and supporting documentation will be evaluated by the study's data-sharing committee. Researchers must submit a proposal detailing their study objectives, statistical analysis plans, and ethical approval. Access will be granted for scientifically valid purposes, following a signed data use agreement. Requests should be directed to: mariagrazia.maggio@irccsme.it.

REFERENCES:
- [Background] Isernia S, Di Tella S, Pagliari C, Jonsdottir J, Castiglioni C, Gindri P, Salza M, Gramigna C, Palumbo G, Molteni F, Baglio F. Effects of an Innovative Telerehabilitation Intervention for People With Parkinson's Disease on Quality of Life, Motor, and Non-motor Abilities. Front Neurol. 2020 Aug 13;11:846. doi: 10.3389/fneur.2020.00846. eCollection 2020. PMID 32903506
- [Background] Barnes DE, Yaffe K, Belfor N, Jagust WJ, DeCarli C, Reed BR, Kramer JH. Computer-based cognitive training for mild cognitive impairment: results from a pilot randomized, controlled trial. Alzheimer Dis Assoc Disord. 2009 Jul-Sep;23(3):205-10. doi: 10.1097/WAD.0b013e31819c6137. PMID 19812460
- [Background] Amjad I, Toor H, Niazi IK, Pervaiz S, Jochumsen M, Shafique M, Haavik H, Ahmed T. Xbox 360 Kinect Cognitive Games Improve Slowness, Complexity of EEG, and Cognitive Functions in Subjects with Mild Cognitive Impairment: A Randomized Control Trial. Games Health J. 2019 Apr;8(2):144-152. doi: 10.1089/g4h.2018.0029. Epub 2018 Sep 21. PMID 30239213